CLINICAL TRIAL: NCT06353295
Title: Community-based, Peer-delivered PrEP for Female Sex Workers in Rural Uganda: The Peers for PrEP (P4P) Study
Acronym: P4P
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of California, San Francisco (Other)
Collaborators: Gilead Sciences (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Prevention
Other Study IDs: 22-38098; CO-US-412-6436 (Other Grant/Funding Number: Gilead Sciences)
Record Dates: First submitted 2024-04-01; First posted 2024-04-09 (Actual); Last update posted 2025-07-14 (Actual); Status verified 2025-07

CONDITIONS: HIV/AIDS
Keywords: Biomedical HIV Prevention; Peer Mentor Intervention; Women Engaged in Sex Work; Uganda
MeSH Terms: conditions — Acquired Immunodeficiency Syndrome

STUDY DESIGN:
Intervention Model Description: A single-arm pilot trial to evaluate a community-based, peer-led and delivered intervention to provide biomedical prevention products (e.g. pre-exposure prophylaxis [PrEP] and post-exposure prophylaxis [PEP]) for women who engage in sex work in southwestern Uganda. This study will test whether the intervention is feasible, acceptable, and increases biomedical prevention uptake.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: Yes

ARMS (1):
- P4P intervention (Other): Peer-led PrEP/PEP intervention
  Interventions: Other: P4P intervention

INTERVENTIONS:
Other: P4P intervention — The final Peers for PrEP (P4P) intervention components were refined based on stakeholder engagement, key informant interviews, and focus group discussions. Trained peers will deliver the following intervention with remote clinician support and ongoing mentorship: pre-exposure prophylaxis (PrEP) access and refills in community/at hotspots; HIV testing, with option for HIV self-testing (HIVST); Rapid post-exposure prophylaxis (PEP) access for unplanned exposures; Family planning integration; Phone/text messaging hotline for peer support

SUMMARY:
The overall goal of the P4P: Peers for PrEP (pre-exposure prophylaxis) study is to pilot test a peer-led and delivered intervention for biomedical HIV prevention that is tailored to women who engage in sex work in southwestern Uganda. This study will evaluate whether this intervention is feasible, acceptable, and increases uptake of biomedical prevention.

DETAILED DESCRIPTION:
The investigators have collaborated with key stakeholders to develop a community-based, peer-led intervention to provide biomedical prevention products (e.g. pre-exposure prophylaxis [PrEP] and post-exposure prophylaxis [PEP]) for women who engage in sex work in southwestern Uganda. A single-arm pilot trial will evaluate the feasibility, acceptability, and preliminary effectiveness of the intervention. The intervention is designed to reduce stigma associated with attending clinics (via community-based delivery by peers), leverage peer support to foster adherence, and reduce barriers to prevention services (through access to PrEP, HIV self-testing, and PEP from trusted peers).

ELIGIBILITY:
Inclusion Criteria:

* Female sex at birth
* Self-identified as commercial sex worker; exchange of sex for goods or money in last 3 months; or work or live in setting associated with sex work
* Age >=18 years (or mature minor >=15 years)
* HIV-negative by country-standard rapid testing algorithm

Exclusion Criteria:

* Contraindication to country-recommended PrEP regimen per national guidelines
* Unable or unwilling to provide informed consent
* Participation in another HIV prevention study

Min Age: 15 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Gender Based: Yes — Female sex at birth
Enrollment: 140 (Estimated)
Dates: Start 2024-04-24 (Actual); Primary Completion 2025-02-14 (Actual); Study Completion 2026-06-30 (Estimated)

PRIMARY OUTCOMES:
Uptake of biomedical prevention | 6 months
  Number of participants receiving biomedical prevention (e.g., oral pre-exposure prophylaxis [PrEP] or post-exposure prophylaxis [PEP]) divided by the number of participants

SECONDARY OUTCOMES:
Feasibility of delivery of the P4P intervention by peers | 6 months
  Feasibility of the P4P intervention will be assessed based on number of participants with services delivered by a peer divided by the number of participants
Acceptability of the P4P intervention | 6 months
  The acceptability of the P4P intervention will be assessed based on participant responses to a post-intervention survey on the acceptability of the intervention

CONTACTS AND LOCATIONS:
Overall Officials: Catherine Koss, MD, Principal Investigator — University of California, San Francisco
Locations (1):
- Infectious Diseases Research Collaboration, Kampala, Uganda

IPD SHARING:
Plan to Share IPD: No